CLINICAL TRIAL: NCT00072891
Title: Improving Medication Adherence in Comorbid Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 59048DK (completed)
Record Dates: First submitted 2003-11-12; First posted 2003-11-14 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemia
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias; Diabetes Mellitus

INTERVENTIONS:
Behavioral: telephone counseling

SUMMARY:
This study is designed to study how adults with Type 2 Diabetes and either high blood pressure and/or high blood cholesterol manage their treatment regimen. It is also called the Diabetes Management Study. Individuals need to be 40 years of age or older and on oral medication (pills) management for two of the three conditions of interest. They may also be on other treatment such as insulin, diet and/or exercise programs. Individuals will be followed for approximately 12 months. About 1/4 of the persons in the study will receive a telephone counseling program with a nurse focused upon their management of their treatment program.

ELIGIBILITY:
* Type 2 diabetes mellitus, hypertension and/or hyperlipidemia,
* On oral medication for two of the above conditions,
* Manage own medications,
* Must have access to a telephone,
* Not participating in other adherence education or counseling trials

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States